CLINICAL TRIAL: NCT02047968
Title: Wake and Light Therapy to In-patients With Major Depression: A Randomized Controlled Trail, Efficacy, Predictors and Patient Experiences
Brief Title: Wake and Light Therapy to In-patients With Major Depression: Efficacy, Predictors and Patient Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VT12
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Major Depression
Keywords: Wake therapy; Sleep deprivation; Light therapy; Bipolar depression; Sleep-wake cycle; Major depression; Depression; Depressive Disorder; Major Behavioural Symptoms; Mood Disorders; Mental Disorders; Dyssomnias; Sleep Disorders; Affective Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Deprivation; Bipolar Disorder; Depression; Depressive Disorder; Mood Disorders; Mental Disorders; Dyssomnias; Sleep Wake Disorders | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wake therapy, light therapy and sleep time stabilisation (Experimental): Wake therapy/sleep deprivation: Patients are awake for 36 hours three times in one week with a normal night of sleep between. Light therapy for 30 minutes daily in the entire study period. Sleep time stabilisation which involves psychoeducation regarding sleep hygiene and keeping the day-night cycle constant.
  Interventions: Behavioral: wake therapy
- treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: wake therapy
  Other Names: light therapy; sleep time stabilisation
  Arms: wake therapy, light therapy and sleep time stabilisation

SUMMARY:
The objective of the study is to examine whether a combination of wake therapy, light therapy and sleep time stabilization as a supplement to standard treatment can reduce depressive symptoms in patients admitted at two psychiatric wards at Aarhus University Hospital, Risskov. Seventy-four patients will be randomized either to this intervention or to a control group receiving treatment as usual. Furthermore, it will be examined whether the duration of admission can be reduced in the intervention group. Finally, the aim is to identify predictors of good effect of the intervention.

DETAILED DESCRIPTION:
Background: About 150,000 Danes will constantly have symptoms of depression, and 20% of those are admitted to a psychiatric hospital at least once. When admitted, the patients are highly tormented and many have suicide thoughts. The treatment of depression in a ward consists of beginning or adjustment of antidepressive medication combined with for instance milieu therapy, psychotherapy and exercise offers. Full effect of medical treatment is only reached after 4-6 weeks, and no quicker effect is documented in the other treatment methods. Therefore, methods are needed which quickly, effectively and without large side effects can reduce the symptoms. Wake therapy is a treatment method which has appeared to stop or reduce depressive symptoms within hours, and several studies have demonstrated that up to 66% of the patients responded to wake therapy. The method consists in the patients staying awake for one night and the following day, in all 36 hours, which is followed by one night of sleep. Light therapy and stabilisation of circadian rhythm have been shown to maintain the effect of wake therapy.

Objective: To examine the efficacy of using wake and light therapy as a supplement to standard treatment of hospitalised patients with depression and to identify the characteristics of patients who accept and respond well to the treatment.

Methods: The project is carried out as a randomised controlled study and will include 74 patients with bipolar or unipolar depression. The patients are randomised to standard treatment or to the intervention, which besides standard treatment will consist of three times wake therapy in one week and 30 minutes daily light treatment in the entire nine week study period as well as ongoing guidance in good sleep hygiene. Raters for the Hamilton rating will be blinded to the treatment assignment.

Outcome: Primary outcome criteria will be the response rate in week two. Response is defined as a 50 % reduction or more compared to the baseline score in HAM-D 17. Secondary outcomes will be the remission rate in week two, the length of admission and the percentage of patients with response and remission in week nine.

Variables and Assessment: Severity of depression will be assessed by using the interview-based Hamilton Depression Rating scale, both the 17 item and the 6 item version. For patient-reported outcome measures the Major Depression Inventory (MDI) and the World Health Organisation (WHO)-5 wellbeing Index (WHO-5) will be used. Social and Occupational Functional Assessment Scale (GAF) and Bech-Rafaelsen mania scala (MAS) will also be recorded.

Data analysis: Data will be analysed in SPSS and presented descriptively in the two Groups to show whether the randomisation succeeded. A "intention to treat" analysis will be conducted, and on the basis of a requisite analysis a t-test, Mann-Whitney-Wilcoxon test or chi2-test will be used. The association between predictive factors and response to wake therapy will be described with prevalence proportions, ratios and will be analysed with a chi2-test. The level of statistical significance will be set at 5 %. The randomisation will be computer-generated, and the patients will be randomly allocated to the intervention group or the control group.

Sample size: The literature shows response rates at 41% after two weeks in the intervention group and 13 % in the control group. A power analysis based on these rates show that if α = 0,05 and β = 0,80, 37 patients should be included in each group, totally 74 patients.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of major depression according to DSM-IV
* A score on the Hamilton Depression Scale, 17 items version of at least 18
* Patient with major depression as part of a bipolar disorder should be in adequate mood stabilising therapy at entry to the study
* Age of 18 to 65
* Speak and understand Danish

Exclusion Criteria:

* Severe suicidal ideation (a score of 3 or above on the Hamilton Depression Scale, 17-items version)
* Anxiety psychic or somatic (a score of 3 or above on the Hamilton Depression Scale, 17-items version)
* personality disorder according to DSM-IV
* Drug or alcohol abuse
* Psychotic disorder
* Pregnancy
* Glaucoma
* Epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Response | Week two
  Response is defined as a 50 % reduction or more compared to the baseline score in HAM-D 17.

SECONDARY OUTCOMES:
Remission | Week two
  Remission will be defined as a score of <8 in HAM-D 17.
Length of admission | Week nine
Percentage of patients with response | week nine
  Response is defined as a 50 % reduction or more compared to the baseline score in HAM-D 17.
Percentage of patients with remission | week nine
  Remission will be defined as a score of <8 in HAM-D 17.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Kragh, RN, MSc, PhDstudent, Principal Investigator — Department of Affective Disorders Q
Locations (1):
- Mette Kragh, Risskov, Central Jutland, Denmark